CLINICAL TRIAL: NCT04272320
Title: The Efficacy of Transversalis Fascia Plane Block on Postoperative Pain in Pediatric Inguinal Hernia Repair
Brief Title: The Efficacy of Transversalis Fascia Plane Block in Pediatric Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Elif Oral Ahiskalioglu, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pediatrik TFP
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (No Intervention)
- Group TFP (Active Comparator): Transversalis fascia plane block, before the surgical procedure.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Ultrasound-guided Transversalis Fascia Plane Block with 0.5 ml/kg %0.25 bupivacaine
  Arms: Group TFP

SUMMARY:
In patients undergoing lower abdominal surgery, postoperative pain management is frequently provided with systemic opioids use or neuraxial methods. Ultrasound-guided TFP block is the preferred method to reduce the use of opioids and systemic analgesics for postoperative pain management. TFP block provides anesthesia and analgesia in the inguinal region by blocking the ilioinguinal and iliohypogastric nerves.

In this study, we aimed to evaluate the effects of ultrasound-guided TFP Block on postoperative pain scores in pediatric lower abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-II patients undergoing ınguinal hernia repair

Exclusion Criteria:

* American Society of Anesthesiologist's physiologic state III-IV

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Pain Score | Postoperative first 24 hours
  Pain will be evaluated with a FLACC (Face, Legs, Activity, Cry, Consolability) score of 0-10 (0= no pain and 10= worst pain)

SECONDARY OUTCOMES:
Additional Analgesic | Postoperative first 24 hours
  Additional Analgesic consumption during postoperative 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Ahiskalioglu A, Aydin ME, Doymus O, Yayik AM, Celik EC. Ultrasound guided transversalis fascia plane block for lower abdominal surgery: First pediatric report. J Clin Anesth. 2019 Aug;55:130-131. doi: 10.1016/j.jclinane.2018.12.046. Epub 2019 Jan 15. No abstract available. PMID 30658324